CLINICAL TRIAL: NCT07245628
Title: A Single-Blind Randomized Placebo Controlled Trial of Self-Adjusted Nitrous Oxide During Office Vasectomy
Brief Title: A Trial of Self-Adjusted Nitrous Versus Placebo During Office Vasectomy
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Alexandra J. Berger Eberhardt, MD (Other)
Responsible Party: Sponsor-Investigator, Alexandra J. Berger Eberhardt, MD, Associate Surgeon, Department of Urology, Brigham and Women's Hospital; Assistant Professor, Harvard Medical School, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025P000258
Record Dates: First submitted 2025-11-10; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Vasectomy
Keywords: Vasectomy; Nitrous Oxide; Men's Health
MeSH Terms: interventions — Nitrous Oxide; Oxygen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nitrous Oxide (Experimental): Self-Administered Nitrous Oxide
  Interventions: Drug: Nitrous Oxide
- Placebo (Oxygen) (Placebo Comparator): Self-Administered Placebo (Oxygen)
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Nitrous Oxide — Self-Administered Nitrous Oxide
  Arms: Nitrous Oxide
Drug: Oxygen — Self-Administered Oxygen
  Arms: Placebo (Oxygen)

SUMMARY:
The goal of this clinical trial is to see if nitrous oxide is safe and effective to use during during vasectomies performed in a clinic/in-office setting.

This trial will compare self-administered nitrous oxide versus a placebo (oxygen) during office vasectomy.

The main questions it aims to answer are:

* Whether self-administered low dose (20-45%) nitrous oxide (SANO) reduces intraoperative anxiety and catastrophizing during office vasectomy.
* To examine whether SANO reduces intraoperative pain or alters procedure duration, the rate of adverse events, or urologists' perception of ease and patient tolerance of the procedure.

Participants will be asked to complete multiple surveys pre-procedure, intra-procedure, and post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 85 at the time of screening
* Desiring vasectomy for family planning purposes
* Able to understand and complete patient questionnaires
* Willing and able to provide written consent to participate in the study

Exclusion Criteria:

* Patients with unilateral absence of the vas deferens
* Patients who are deemed by study surgeons to have anatomy no amendable for office procedure
* Patients who decline office vasectomy and request monitored anesthesia care
* Patients taking benzodiazepine or narcotic medication daily or within 24 hours of the procedure
* Patients with contraindications to nitrous oxide including:
* Inner ear, bariatric, or eye surgery within the past 2 weeks
* Current emphysematous blebs
* Severe B-12 deficiency
* History of bleomycin chemotherapy within the last year
* Class III or higher heart failure

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
Mean Difference in VAS-A During Vasectomy Procedure and S-PCS Immediately After Vasectomy Procedure, Comparing Participants Receiving and Not Receiving Self-Administered Low Dose Nitrous Oxide | Intra-Procedure (Immediately After Injection of Local Anesthesia) - Post-Procedure (10 Minutes After Procedure Completion, Allow for Nitrous Oxide to be Metabolized)
  Measuring the mean difference in Visual Analog Scale for Anxiety (VAS-A) during the vasectomy procedure and the Situational Pain Catastrophizing Scale (S-PCS) immediately after the vasectomy procedure, comparing those receiving and not receiving self-administered low dose nitrous oxide.
  Intra-Procedure (Immediately After Injection of Local Anesthesia) Visual Analog Scale for Anxiety (VAS-A) (Zero is equivalent to no anxiety and 10 indicates the worst anxiety)
  Intra-Procedure (In Between Left and Right Sides of Procedure) Visual Analog Scale for Anxiety (VAS-A) (Zero is equivalent to no anxiety and 10 indicates the worst anxiety)
  Post-Procedure (10 Minutes After Procedure Completion, to Allow for Nitrous Oxide to be Metabolized)
  1. Situational Pain Catastrophizing Scale (S-PCS) (Zero is equivalent to not at all and 4 indicates all the time)
  2. Visual Analog Scale for Anxiety (VAS-A) (Zero is equivalent to no anxiety and 10 indicates the worst anxiety)

SECONDARY OUTCOMES:
Mean Difference in Visual Analog Scale for Pain (VAS-P) Intra-Procedurally, Comparing Participants Receiving and Not Receiving Self-Administered Low Dose Nitrous Oxide | Intra-Procedure (Immediately After Injection of Local Anesthesia) - Intra-Procedure (In Between Left and Right Sides of Procedure)
  Intra-Procedure (Immediately After Injection of Local Anesthesia) Visual Analog Scale for Pain (VAS-P) (Zero is equivalent to no pain and 10 indicates the worst pain)
  Intra-Procedure (In Between Left and Right Sides of Procedure) Visual Analog Scale for Pain (VAS-P) (Zero is equivalent to no pain and 10 indicates the worst pain)
Mean Difference in VAS-P and STAI Pre- and Post-Procedurally, Comparing Participants Receiving and Not Receiving Self-Administered Low Dose Nitrous Oxide | Pre-Procedure (Day of Procedure, Immediately Prior) - Post-Procedure (10 Minutes After Procedure Completion, Allow for Nitrous Oxide to be Metabolized)
  Pre-Procedure (Day of Procedure, Immediately Prior)
  1. Visual Analog Scale for Pain (VAS-P) (Zero is equivalent to no pain and 10 indicates the worst pain)
  2. State Trait Anxiety Inventory (STAI) (1 is equivalent to not at all and 4 indicates very much)
  Post-Procedure (10 Minutes After Procedure Completion, Allow for Nitrous Oxide to be Metabolized)
  1. Visual Analog Scale for Pain (VAS-P) (Zero is equivalent to no pain and 10 indicates the worst pain)
  2. State Trait Anxiety Inventory (STAI) (1 is equivalent to not at all and 4 indicates very much)
Mean Difference in 30-Day Complications / Adverse Events, Comparing Participants Receiving and Not Receiving Self-Administered Low Dose Nitrous Oxide | Study Enrollment - 30 Days After Vasectomy
  Measured using the The Common Terminology Criteria for Adverse Events (CTCAE) grading scale (v5.0).
  CTCAE v5.0 (1 is equivalent to mild and 5 indicates death related to AE)
Urologist: Ease of Procedure, Comparing Participants Receiving and Not Receiving Self-Administered Low Dose Nitrous Oxide | Post-Procedure, Day of Vasectomy
  Post-Procedure, Day of Vasectomy Ease of Procedure (1 is equivalent to the urologist determining the procedure went worse than expected and 3 indicates the urologist determines the procedure went better than expected)
Urologist: Patient Tolerance, Comparing Participants Receiving and Not Receiving Self-Administered Low Dose Nitrous Oxide | Post-Procedure, Day of Vasectomy
  Patient Tolerance (1 is equivalent to the urologist determining the patient's tolerance for the procedure was worse than expected and 3 indicates the urologist determines the patient's tolerance for the procedure was better than expected)
Mean Difference in Duration of Procedure, Comparing Participants Receiving and Not Receiving Self-Administered Low Dose Nitrous Oxide | Intra-Procedure (Immediately After Injection of Local Anesthesia) - Post-Procedure (10 Minutes After Procedure Completion, Allow for Nitrous Oxide to be Metabolized)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra J Berger Eberheardt, MD, Study Chair — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes